CLINICAL TRIAL: NCT06813625
Title: Shared Book Reading to Promote Mental Well-being Among Young People with and Without Down's Syndrome: a Pilot Dyadic Randomized Controlled Trial
Brief Title: Shared Book Reading to Promote Mental Well-being Among Young People with and Without Down's Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Macau (Other)
Responsible Party: Principal Investigator, Robert Smith, Assistant Professor, University of Macau
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HE-0442-2025
Record Dates: First submitted 2025-01-27; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shared book reading intervention (Experimental): An 8-week pilot binary randomized controlled trial involving one hour of shared book reading per week in young people with and without Down syndrome.
  Interventions: Behavioral: Shared book reading intervention
- Control Group (No Intervention): Those in the control group will be informed that they will wait 8 weeks before they can join the shared book reading sessions. Dyads will not be put in contact with each other. To keep young people with DS engaged with the study, those in the control group will be offered 3 books, from the selection of 20, that they can read themselves during the control period. After the 8-week period those that attend the shared book reading sessions will be introduced to their dyadic partner to participate in the sessions fully.

INTERVENTIONS:
Behavioral: Shared book reading intervention — The intervention involved us pairing each teen DS with a college student to form a duo. Each group consists of one person with DS and at least one college student who will work together throughout the shared reading intervention. A weekly event hosted by a graduate student. It begins with ice-breaking activities such as color and music games to promote social interaction between participants. After the game, participants chose from a selection of 20 books suitable for different age groups. They can choose their own reading method, such as reading aloud or assigning roles, and are encouraged to share experiences in their own duos or in a large group of multiple duos. The session ends with a sharing and reflection activity where participants can discuss what they have read and plan for the next session.
  Arms: Shared book reading intervention

SUMMARY:
Abstract Background: With the progress of society and the deepening of people's understanding of Down syndrome (DS), research has shifted focus on how to improve the quality of life and education for young people with DS. This study shall pilot a shared book reading intervention to test for potential benefit and feasibility.

Methods: This study is an 8 weeks long pilot dyadic randomized controlled trial (RCT) comparing a shared book reading intervention to a minimal activity control, this study will then continue for 12 months as a single arm cohort study. Young people with DS and university undergraduate students will be recruited and formed into dyads then randomized to either intervention or control. The shared book reading activity will include partnering young people with DS and university students together for a weekly, 1-hour shared book reading session. The control group will be supplied with three books they can read in their free time during 8 weeks. The primary outcomes included young people with DS health-related quality of life measured using the Children's Quality of Life Scale (PedsQL4.0). Secondary outcomes include mental well-being in university students using the Engagement, Perseverance, Optimism, Connectedness, and Happiness scale (EPOCH). Measurements will be made at baseline (T0) and 8-week (T1). After 8 weeks all participants will be offered to continue in the study where all participants will join the shared book reading weekly intervention and outcomes measures will be made at 6-month (T2), and 12-month (T3) follow-up. Mixed linear regression models shall be conducted comparing intervention and control group at 8 weeks. At 6-months and 12-months follow-up change scores from baseline will be analyzed to test for potential long-term effect.

Anticipated results: If our pilot study can show that shared book reading activities for people with DS can be of benefit and feasible, this can lead to a fully powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria for Participants with Down Syndrome (DS):

* Clinical diagnosis of Down Syndrome (DS).
* Aged 2 years or older.
* Able to participate in the intervention and study evaluation independently or with the support of caregivers or family members.

Inclusion Criteria for University of Macau (UM) Students:

* Aged 18 years or older.
* Able to read and understand books in English or Chinese.
* Able to communicate in English, Mandarin, or Cantonese.
* Do not have severe visual or reading disabilities that may affect reading ability.

Exclusion Criteria:

-Have severe visual or reading disabilities.

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-08 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
PedsQL4.0 | PEDSQL4.0 is assessed at three time points: Baseline (T0), 8 weeks (T1), and 6 months (T2). This allows for tracking changes in health-related quality of life over time among participants.
  Health related quality of life for young people with DS will be measured using the Children's Quality of Life Scale (PedsQL4.0). The Child Quality of Life Scale (PedsQL) is a common tool used to assess a child's quality of life and can be used to measure quality of life (QOL) in children and adolescents aged 2-18 years with acute or chronic medical conditions, including DS. The PedsQL4.0 covering domains of physical functioning, emotional state, social interaction, and school performance, as well as providing a total score for overall quality of life. The PedsQL4.0 items ask to what extent the participant has had problems in the past month. The higher the score on the PedsQL4.0 tool indicates a higher the quality of life. The questionnaire showed good psychometric characteristics among young people and internal consistency (Cronbach's alpha range was 0.66 to 0.93).

SECONDARY OUTCOMES:
The Global Perceived Effects scale (GPE) | GPE is assessed at this time points: 8 weeks (T1). This allows for tracking changes in health-related quality of life over time among participants.
  The Global Perceived Effects scale (GPE) used in the responsiveness analysis and for determining the minimal important change. Caregivers choosing response options"very much improved"and"much improved"were considered to have "importantly improved,"and those choosing options 3-5 ("a little improved, no change and a little deterioration") were considered to be"stable."For research or clinical evaluation to understand the impact of shared book reading activities on children's quality of life and their caregivers. This information is valuable to doctors, researchers, and healthcare providers because it can help them evaluate the effects of interventions and improve future intervention strategies.
EPOCH | EPOCH is assessed at three time points: Baseline (T0), 8 weeks (T1), and 6 months (T2). This allows for tracking changes in mental health over time among participants.
  The EPOCH Measure of Adolescent Well-being is a scale used to assess positive psychological traits in adolescents. It consists of 20 items with five dimensions: Engagement, Perseverance, Optimism, Connectedness and Happiness. This scale was developed to assess five positive psychological traits that may promote well-being, physical health, and other positive outcomes in adulthood. The scale is an effective tool that provides a short and reliable measurement tool for schools or organizations to help assess a youth's sense of psychological well-being.
  * Score Range: Typical Likert-type scales (e.g., 1-5 or 0-4) are often used, so the total score range would depend on the response format (e.g., 20-100 if a 1-5 scale is used).
  * Interpretation: Higher scores indicate better outcomes (i.e., greater psychological well-being).
Friendship quality questionnaire (FQQ) | FQQ is assessed at time points: 6 months (T2). This allows for tracking changes in friendship quality over time among participants.
  Friendship Quality Questionnaire (FQQ)
  * Purpose: Assesses the quality of friendship among children and adolescents across five dimensions.
  * Dimensions: Companionship、Conflict、Helpfulness、Security and Closeness.
  * Score Range: If the questionnaire uses a Likert-type scale (e.g., 1-5 or 0-4), the total score range would depend on the number of items and response options.
  * Interpretation: Higher scores indicate better outcomes (i.e., higher quality of friendship).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Macau, Macau, China

IPD SHARING:
Plan to Share IPD: Undecided
Due to the small number of children with Down's syndrome in Macau SAR and the scope of this study, anonymized individual data may become identifiable.

REFERENCES:
- [Background] Perra A, Primavera D, Leonetti V, Montisci R, Carta D, Lorrai G, Locci A, Chessa L, Scuteri A, Cossu G, Nardi AE, Valmaggia L, Galetti A, De Lorenzo V, Sancassiani F, Carta MG. Virtual reality cognitive remediation tool for individuals with mild cognitive impairment: study protocol for a feasibility randomized clinical trial. Front Public Health. 2024 Nov 22;12:1477279. doi: 10.3389/fpubh.2024.1477279. eCollection 2024. PMID 39651467
- [Background] Peiris DLIHK, Duan Y, Vandelanotte C, Liang W, Baker JS. In-classroom physical activity breaks program among school children in Sri Lanka: study protocol for a randomized controlled trial. Front Public Health. 2024 Apr 22;12:1360210. doi: 10.3389/fpubh.2024.1360210. eCollection 2024. PMID 38711768
- [Background] Bridi D, Valentini NC, Deslandes AC, Copetti F. Focused attention and intrinsic motivation using animations for instruction of fundamental motor skills in children with Down syndrome. J Intellect Disabil Res. 2024 Aug;68(8):954-968. doi: 10.1111/jir.13140. Epub 2024 Apr 21. PMID 38644604
- [Background] Hsu CF, Jiang Q, Rao SY. Category-Based Effect on False Memory of People with Down Syndrome. Brain Sci. 2024 May 24;14(6):538. doi: 10.3390/brainsci14060538. PMID 38928536
- [Background] Grover V, Snow CE, Evans L, Stromme H. Overlooked advantages of interactive book reading in early childhood? A systematic review and research agenda. Acta Psychol (Amst). 2023 Sep;239:103997. doi: 10.1016/j.actpsy.2023.103997. Epub 2023 Aug 8. PMID 37562321
- [Background] Frizelle P, O'Donovan S, Jolley M, Martin L, Hart N. The co-construction of a reading assessment measure with adults with Down syndrome: a meaningful literacy approach. Front Psychol. 2023 Jul 20;14:1173300. doi: 10.3389/fpsyg.2023.1173300. eCollection 2023. PMID 37546441
- [Background] Dong Y, Mo J, Gong B, Jin R, Zheng H, Chow BW. Effects of Using Prompts During Parent-Child Shared Reading on the Language Development of Mildly Autistic Children. J Autism Dev Disord. 2025 Jan 11. doi: 10.1007/s10803-024-06712-9. Online ahead of print. PMID 39797957
- [Background] Akkarakittichoke N, Janwantanakul P, Kanlayanaphotporn R, Jensen MP. Responsiveness of the UW Concerns About Pain Scale and UW Pain-Related Self-Efficacy Scale in Individuals With Chronic Low Back Pain. Clin J Pain. 2022 Jul 1;38(7):476-483. doi: 10.1097/AJP.0000000000001043. PMID 35686577
- [Background] Wiwaha G, Sari DM, Biben V, Sunjaya DK, Hilmanto D. Translation and validation of Indonesian version of Pediatric Quality of Life Inventory (PedsQL) Neuromuscular Module. Health Qual Life Outcomes. 2022 Feb 24;20(1):33. doi: 10.1186/s12955-022-01933-x. PMID 35209927
- [Background] Kamdem F, Meyanga Ngoah J, Nganou Gnindjio CN, Mekoulou Ndongo J, Ba H, Mouliom S, Viche L, Ngote H, Kenmegne C, Tsague Kengni H, Ndom Ebongue MS, Djibrilla S, Bika Lele EC. Pattern and determinants of health-related quality of life of adolescents with congenital heart disease in Cameroon: A single-center cross-sectional study. JRSM Cardiovasc Dis. 2024 Apr 17;13:20480040241247396. doi: 10.1177/20480040241247396. eCollection 2024 Jan-Dec. PMID 38638397
- [Background] Guevara VLS, Coelho RF, Flores EP. Effects of dialogic reading for comprehension (LuDiCa) on the social interaction of autistic adolescents and their peers. Psicol Reflex Crit. 2024 Feb 2;37(1):4. doi: 10.1186/s41155-023-00283-x. PMID 38305847
- [Background] Na JY, Wilkinson KM. Communication about emotions during storybook reading: Effects of an instruction programme for children with Down syndrome. Int J Speech Lang Pathol. 2018 Dec;20(7):745-755. doi: 10.1080/17549507.2017.1356376. Epub 2017 Aug 7. PMID 28780903
- [Background] Munoz-Llerena A, Ladron-de-Guevara L, Medina-Rebollo D, Alcaraz-Rodriguez V. Impact of Physical Activity on Autonomy and Quality of Life in Individuals with Down Syndrome: A Systematic Review. Healthcare (Basel). 2024 Jan 11;12(2):181. doi: 10.3390/healthcare12020181. PMID 38255069
- [Background] Neitzel I. Narrative abilities in individuals with Down syndrome: single case-profiles. Front Psychol. 2023 Oct 3;14:1116567. doi: 10.3389/fpsyg.2023.1116567. eCollection 2023. PMID 37854146
- [Background] Alqahtani AS, Algabbani MF, Alhammad SA, Alwadeai KS, Alhusaini A. Physical activity status and its association with quality of life among children with down syndrome in Saudi Arabia: A comparative cross-sectional study. PLoS One. 2024 Feb 12;19(2):e0297111. doi: 10.1371/journal.pone.0297111. eCollection 2024. PMID 38346033
- [Background] Long KL, Karimi A, Mini A, Stephens DP, Nelson EL. The meaning of adulthood for emerging adults with Down syndrome: Parent perspectives on relevant skills. J Appl Res Intellect Disabil. 2024 Sep;37(5):e13286. doi: 10.1111/jar.13286. PMID 39075798
- [Background] Hosseini SJ, Ramezani M, Ashrafzadeh F, Jamali J. Motivation in caregiving among mothers of children with intellectual and developmental disabilities in Iran: A qualitative study. BMC Pediatr. 2024 Jul 25;24(1):472. doi: 10.1186/s12887-024-04957-y. PMID 39049077
- [Background] Burgoyne K, Pagnamenta E, Hartwell K, Stojanovik V. Protocol for a randomised controlled feasibility trial of parent-delivered early language intervention for children with Down syndrome (PACT-DS). Pilot Feasibility Stud. 2023 Dec 7;9(1):196. doi: 10.1186/s40814-023-01419-7. PMID 38062458
- [Background] van Gameren-Oosterom HB, Buitendijk SE, Bilardo CM, van der Pal-de Bruin KM, Van Wouwe JP, Mohangoo AD. Unchanged prevalence of Down syndrome in the Netherlands: results from an 11-year nationwide birth cohort. Prenat Diagn. 2012 Nov;32(11):1035-40. doi: 10.1002/pd.3951. Epub 2012 Aug 6. PMID 22865545
- [Background] Mannion A, Neil N, Fiani T, Athamanah L, Lyons J, McDonagh K, Boland E, Cooney R, Lynch M, Youssef M, Leader G. An investigation of sleep problems, gastrointestinal symptoms, comorbid psychopathology and challenging behavior in children and adolescents with Down Syndrome. Res Dev Disabil. 2024 Aug;151:104788. doi: 10.1016/j.ridd.2024.104788. Epub 2024 Jul 3. PMID 38964213
- [Derived] Huang X, Long I, Zhang W, Xu J, Smith RD. Shared book reading to promote mental well-being among young people with and without Down syndrome: a pilot dyadic randomized controlled trial. Front Public Health. 2025 Oct 29;13:1604241. doi: 10.3389/fpubh.2025.1604241. eCollection 2025. PMID 41235213